CLINICAL TRIAL: NCT01371929
Title: Evaluation of the PliNOSa® Test as an Aid in the Risk Assessment for the Onset of Sepsis
Brief Title: Plasma Inducible Nitric Oxide Synthase (iNOS) Assay and Sepsis Study
Acronym: PliNOSa® Test
Status: Terminated | Type: Observational
Why Stopped: NIH funding ended prior to full enrollment in the clinical study
Sponsor: Research & Diagnostic Antibodies (Industry)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Dr. Robert Webber, President, Research & Diagnostic Antibodies
Other Study IDs: RDAbs 11-001; 1RC3GM093717-01 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-06-13 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — heparinized plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ICU patients who become septic: Patients considered to be at risk of becoming septic based upon his/her clinical presentation during admittance or transfer to an ICU will be tested for the presence of plasma iNOS using our PliNOSa test on the day of ICU entry and their sepsis status will be followed for three days to determine if they develop sepsis, severe sepsis, or septic shock. Approximately, 50% of the enrolled patients are expected to develop sepsis, severe sepsis, or septic shock.
- ICU patients who do not become septic: Patients considered to be at risk of becoming septic based upon his/her clinical presentation during admittance or transfer to an ICU will be tested for the presence of plasma iNOS using our PliNOSa test on the day of ICU entry and their sepsis status will be followed for three days to determine if they develop sepsis, severe sepsis, or septic shock. Approximately, 50% of the enrolled patients are expected NOT to develop sepsis, severe sepsis, or septic shock.

SUMMARY:
The primary objective is to demonstrate that the plasma inducible nitric oxide synthase (iNOS) assay (PliNOSa® test) has an acceptable relative risk ratio for predicting the onset of sepsis within 72 hours of testing when performed on the first day a patient is admitted or transferred to the intensive care unit (ICU) and is considered to be at risk of becoming septic. The PliNOSa® test measures inducible nitric oxide synthase (iNOS) in plasma and uses a pre-determined iNOS cut-off value to identify patients at risk for the onset of the sepsis pathology.

DETAILED DESCRIPTION:
At present, an accurate and definitive clinical test to predict early the onset of the sepsis pathology does not exist. At least 7 million people per year enter into the early stages of the sepsis pathology, which will lead to more than 250,000 deaths per year in the USA and more than 750,000 worldwide. An early, accurate, and reliable test that can assess an intensive care unit (ICU) patient's risk of becoming septic would be a major medical breakthrough. A large unmet clinical laboratory need exists for a test that can aid physicians in assessing their patient's risk for the onset of the sepsis pathology. The current culture procedures suffer from a number of problems. (1) They are slow. The first answer is obtained only after 24 hours of culture, and an absolute answer requires a minimum of 48 hours of culture. (2) Blood culture only yields positive results (i.e. sepsis is present) in approximately 28% of patients who become septic, thus over 70% of the patients do not yield positive blood cultures. Everyone in the sepsis field agrees that better IVD tests for the sepsis pathology are desperately needed. Our PliNOSa IVD test based upon the presence of iNOS in plasma should identify those patients as being at risk for developing sepsis since our assay is not dependent upon the culturing of live bacteria or other micro-organisms.

Sepsis develops from a variety of bacterial and fungal sources stemming from the patient's inability to fight infection, and is commonly acquired while recovering from severe injuries and surgery in hospitals. An early, accurate, and reliable clinical diagnostics test for the onset of sepsis currently does not exist, but an enormous clinical laboratory need does exist. In January 2008, Levenson reviewed the current status of the clinical diagnosis of sepsis and concluded [1] that none of the currently FDA cleared risk-assessment tests work well and [2] that new biomarkers specific for the sepsis pathology would be a major medical breakthrough. In 2000, the Institute of Medicine of the National Academy of Science estimated the cost to the US healthcare system to be $17 - 29 billion annually. The presence in plasma of a normally intracellular protein, inducible nitric oxide synthase (iNOS), has been found to be an early and accurate biomarker for the onset of the sepsis pathology. Data gathered using our in vitro diagnostic (IVD) test to analyze more than 1,200 blood samples collected during our clinical studies on 350 study subjects (295 ICU patients and 55 healthy volunteers) demonstrated that iNOS is present only in plasma samples obtained from people suffering from the onset of sepsis. In our three clinical studies, the latter two of which were partially funded by the NIH, our candidate IVD test for plasma iNOS was found to predict the onset of sepsis 24 - 72 hours before the appearance of the physiological symptoms of the pathology.

The superiority of plasma iNOS as compared to other potential biochemical markers of SIRS (pre-sepsis) and sepsis was assessed using the data from our third clinical study. Four cohorts from this study were analyzed for the plasma levels for four potential biomarkers of the sepsis pathology: iNOS, procalcitonin (PCT), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNFα). The four cohorts are (1) 36 normal healthy individuals as Group A; (2) critically injured patients who remained SIRS and septic negative throughout the entire study period as Group B; (3) critically ill patients who became septic during the study period, with their plasma levels 24 hours before the symptoms of sepsis were recognized by the attending doctors as Group C; and (4) confirmed septic patients who were enrolled in our study and had not received antibiotics prior to their enrollment as Group D. Only plasma iNOS was found to differentiate between non-septic critically ill patients (Group B) and the critically ill patients who were developing sepsis (Group C) or were already septic (Group D). The plasma level of procalcitonin, one of the FDA cleared IVD tests, was not specific for sepsis since a number of normal healthy volunteers and many of the non-SIRS and non-septic patients had elevated plasma levels of procalcitonin (PCT).

To summarize, infections in intensive care units and other hospital settings can be caused by different types of organisms, such as bacteria and fungi. These infections annually cause more than 7,000,000 cases of SIRS (pre-sepsis) that can deteriorate to sepsis, severe sepsis with organ dysfunction, and septic shock with multiple organ failure. To date, three clinical studies have been conducted on this project in which 295 ICU patients and 55 healthy volunteers have been enrolled and studied. The data obtained during these prior clinical studies clearly demonstrate that a measurable increase in the plasma level of iNOS occurs during the onset of the sepsis pathology. The main focus of this research proposal is to gather the data needed to obtain FDA clearance to market our new PliNOSa® test by demonstrating in a statistically significant number of critically ill ICU patients that the presence of iNOS in plasma is a reliable early biomarker as a risk assessment aid for the onset of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* May be designated Do Not Attempt to Resuscitate / Do Not Intubate (DNAR / DNI) if they are committed to FULL CARE
* Study subject or their legal representative must have read, understood and provided written informed consent after the clinical study has been fully explained and their questions answered
* Subject must be admitted to or transferred to an Intensive Care Unit (ICU) and expected to require ICU-level of Care >24 hours for any of the following reasons:

  * Following a surgical procedure
  * Following a traumatic injury
  * For threatened or actual respiratory failure
  * For hemodynamic instability
* Subject is considered to be at risk of developing sepsis during the next 72 hours based upon his/her clinical presentation
* Must have an in-dwelling line from which blood can be drawn.

Exclusion Criteria:

* Cannot be already septic, severely septic or in septic shock as defined by a recent positive culture (< 48 hrs) plus 2 or more of the signs and symptoms of sepsis listed in Table 1, "Diagnostic Criteria for Sepsis" in Levy MM, et al (2003) Crit Care Med, 31#4:1250-1256.
* Cannot be moribund (not expected to survive 48 hours)
* Cannot be expected to be discharged from the ICU in under 3 days
* Cannot be pregnant
* Cannot be a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 290 consecutively enrolled critically ill ICU patients who are considered to be at risk of becoming septic based upon their clinical presentation due to trauma, or a surgical procedure, or threatened or actual respiratory failure, or hemodynamic instability; and recruited from three clinical sites. The first 40 study subjects will comprise the pilot cohort and the remaining 250 study subjects will comprise the pivotal cohort.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the PliNOSa test for a Positive Percent Agreement greater than 75% or a Negative Percent Agreement greater than 75% for predicting in ICU patients the onset of sepsis diagnosed within 72 hours of a plasma sample collected on study day 1. | First 72 hours after entry into the ICU
  A successful result (rejection of the null hypothesis) will be achieved if the Positive Percent Agreement is greater than 75% or the Negative Percent Agreement is greater than 75%.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Webber, Ph.D., Principal Investigator — Research & Diagnostic Antibodies

REFERENCES:
- [Background] Webber RJ, Sweet RM, Webber DS. Inducible Nitric Oxide Synthase in Circulating Microvesicles: Discovery, Evolution, and Evidence as a Novel Biomarker and the Probable Causative Agent for Sepsis. J Appl Lab Med. 2019 Jan;3(4):698-711. doi: 10.1373/jalm.2018.026377. PMID 30937423
- [Background] Webber RJ, Rodriguez JG, Webber DS, Dunnebacke TH. Development, characterization, and epitope mapping of a panel of twenty-four monoclonal antibodies specific for human inducible nitric oxide synthase. Hybridoma (Larchmt). 2005 Feb;24(1):6-13. doi: 10.1089/hyb.2005.24.6. PMID 15785204
- [Background] Sands KE, Bates DW, Lanken PN, Graman PS, Hibberd PL, Kahn KL, Parsonnet J, Panzer R, Orav EJ, Snydman DR, Black E, Schwartz JS, Moore R, Johnson BL Jr, Platt R; Academic Medical Center Consortium Sepsis Project Working Group. Epidemiology of sepsis syndrome in 8 academic medical centers. JAMA. 1997 Jul 16;278(3):234-40. PMID 9218672
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Background] Gambim MH, do Carmo Ade O, Marti L, Verissimo-Filho S, Lopes LR, Janiszewski M. Platelet-derived exosomes induce endothelial cell apoptosis through peroxynitrite generation: experimental evidence for a novel mechanism of septic vascular dysfunction. Crit Care. 2007;11(5):R107. doi: 10.1186/cc6133. PMID 17894858
- [Background] Azevedo LC, Janiszewski M, Pontieri V, Pedro Mde A, Bassi E, Tucci PJ, Laurindo FR. Platelet-derived exosomes from septic shock patients induce myocardial dysfunction. Crit Care. 2007;11(6):R120. doi: 10.1186/cc6176. PMID 17996049
- [Background] Mortaza S, Martinez MC, Baron-Menguy C, Burban M, de la Bourdonnaye M, Fizanne L, Pierrot M, Cales P, Henrion D, Andriantsitohaina R, Mercat A, Asfar P, Meziani F. Detrimental hemodynamic and inflammatory effects of microparticles originating from septic rats. Crit Care Med. 2009 Jun;37(6):2045-50. doi: 10.1097/CCM.0b013e3181a00629. PMID 19384196
- [Background] Marshall JC. Why have clinical trials in sepsis failed? Trends Mol Med. 2014 Apr;20(4):195-203. doi: 10.1016/j.molmed.2014.01.007. Epub 2014 Feb 24. PMID 24581450
- [Background] Tse MT. Trial watch: Sepsis study failure highlights need for trial design rethink. Nat Rev Drug Discov. 2013 May;12(5):334. doi: 10.1038/nrd4016. No abstract available. PMID 23629495